CLINICAL TRIAL: NCT03323476
Title: Maintaining or Stopping Immunosuppressive Therapy in Patients With ANCA Vasculitis and End-stage Renal Disease: a Prospective, Multicenter, Randomized, Open-label, Clinical Trial
Brief Title: Maintaining or Stopping Immunosuppressive Therapy in Patients With ANCA Vasculitis and End-stage Renal Disease
Acronym: MASTER-ANCA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHD005-17
Record Dates: First submitted 2017-10-13; First posted 2017-10-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-11

CONDITIONS: Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; End Stage Renal Disease
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Kidney Failure, Chronic | interventions — Immunosuppression Therapy; Maintenance; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discontinuation of maintenance treatment (Experimental)
  Interventions: Other: Discontinuation (or not initiation) of Immunosuppressive Therapy
- Maintenance of immunosuppressive treatment (Active Comparator)
  Interventions: Drug: Maintenance (or initiation) of immunosuppressive treatment: Imurel®, Mabthera®,Cellcept®, Cortancyl®

INTERVENTIONS:
Other: Discontinuation (or not initiation) of Immunosuppressive Therapy — Discontinuation (or not initiation) of Immunosuppressive Therapy
  Arms: Discontinuation of maintenance treatment
Drug: Maintenance (or initiation) of immunosuppressive treatment: Imurel®, Mabthera®,Cellcept®, Cortancyl® — Maintenance (or initiation) of Immunosuppressive Therapy: Imurel®, Mabthera®,Cellcept®, Cortancyl®
  Arms: Maintenance of immunosuppressive treatment

SUMMARY:
This prospective randomized trial aims to evaluate the feasibility, risk and benefit of the discontinuation of immunosuppressive maintenance treatments in AAV (Antineutrophil Cytoplasmic Autoantibodies (ANCA)-associated vasculitis) patients who have reached ESRD (end-stage renal disease). Our hypothesis is that discontinuation of immunosuppressive therapy in AAV patients with ESRD will not expose these patients to an excessive risk of extra-renal AAV relapse, while reducing the rate of complications due to immunosuppression, particularly infections.

Patients with ESRD related to AAV will be randomized into 2 arms:

arm 1: discontinuation (or not initiation) of maintenance treatment (Experimental group) arm 2: maintenance (or initiation) of immunosuppressive treatment (Control group).

The main objective of this study is to demonstrate a superiority of immunosuppression discontinuation in ESRD-AAV patients compared to standard maintenance immunosuppressive therapy in terms of severe prejudicial event-free survival at 24 months. The second objectives include the frequency of major and minor relapses, of infectious episodes and leukopenia in both groups and the establishment of a prospective database regarding the outcome of ESRD-AAV patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 90 years
* Patients affected by a GPA or MPA AAV with a renal injury
* Patients with initial manifestation or relapse of AAV
* Patients with ESRD, defined by a glomerular filtration rate estimated using the MDRD formula ≤15 mL/min or requirement for dialysis for more than 60 days
* Patients with ESRD on native kidney
* Patients who gave written informed consent for participation in the study
* Patients with affiliation to the French social security system

Exclusion Criteria:

* Patients who experienced severe extra-renal disease due to AAV (intra-alveolar haemorrhage with blood oxygen saturation ≤ 85% on room air or ventilated, or central nervous system disease) in the last 12 months prior to inclusion
* Patients with AAV-associated renal involvement (with active inflammatory lesions in kidney biopsy) diagnosed less than three months and receiving induction treatment with cyclophosphamide or rituximab or diagnosed less than 45 days for patients who have receveid only treatment based on steroid infusion without cyclophosphamide or rituximab
* Patients who received maintenance immunosuppressive treatment for more than 6 months during the last 12 months
* Patient with a diagnosis of vasculitis other than GPA or MPA
* Patients with another immunologic systemic disease (Lupus, sarcoidosis…) Patients with active HCV, HBV or HIV infection
* Patients with a history of serious viral infection (CMV, HHV8, etc.) in the 2 months prior to the inclusion, or severe uncontrolled chronic infection (tuberculosis, etc.)
* Patients with uncontrolled cancer or hemopathy
* Kidney transplant patient
* Inability to understand and sign the informed consent
* Pregnant women.
* Women of child-bearing age without effective method of contraception
* Age < 18 years or > 90 years.
* Patients under guardianship or trusteeship.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2018-02-02 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
The primary end point will be the time between inclusion and the first severe prejudicial event (measured in days) during 24 months of follow-up. | During the 24 months of follow-up
  Severe prejudicial event is defined by the occurrence of: severe infection, major AAV relapse, death

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire COUVRAT-DESVERGNES, Principal Investigator — CHD Vendée
Locations (58):
- France (58):
  - Centre Hospitalier Universitaire Amiens, Amiens
  - CHU Angers, Angers
  - Centre Hospitalier Angoulême, Angoulême
  - Centre Hospitalier ARRAS, Arras
  - Centre Hospitalier Avignon, Avignon
  - AUB Santé, Avranches
  - CHRU Besançon, Besançon
  - Centre Hospitalier Universitaire Bordeaux, Bordeaux
  - APHP Ambroise Paré, Boulogne-Billancourt
  - Centre Hospitalier Boulogne sur Mer, Boulogne-sur-Mer
  - Centre Hospitalier Jacques Coeur, Bourges
  - Centre Hospitalier Universitaire de Brest, Brest
  - Centre Hospitalier René Dubois - Pontoise, Cergy-Pontoise
  - Centre Hospitalier Chartres, Chartres
  - Centre Hospitalier Universitaire G. Montpied, Clermont-Ferrand
  - Hopital Louis Pasteur, Colmar
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - CHI Eure Seine, Évreux
  - Centre Hospitalier Universitaire Grenoble, Grenoble
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Centre Hospitalier La Rochelle, La Rochelle
  - Centre ECHO - Le Mans, Le Mans
  - Centre Hospitalier Le Mans, Le Mans
  - Centre Hospitalier Emile ROUX, Le Puy-en-Velay
  - Hôpital Privé La Louvière, Lille
  - CHRU Lille, Lille
  - Centre Hospitalier Universitaire Dupuytren, Limoges
  - AUB Santé - Lorient, Lorient
  - Centre Hospitalier Lyon Sud, Lyon
  - Hopital de la Conception - APHM, Marseille
  - Centre Hospitalier de Mont de Marsan, Mont-de-Marsan
  - Centre Hospitalier Universitaire Lapeyronie, Montpellier
  - GHR Mulhouse Sud Alsace, Mulhouse
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Centre Hospitalier Universitaire Nice, Nice
  - CHU de Nimes, Nîmes
  - Aphp - Bichat, Paris
  - Aphp - Hegp, Paris
  - APHP - Henri Mondor, Paris
  - CHU Kremlin - Bicêtre, Paris
  - Hôpital Saint Louis, Paris
  - Hôpital Tenon, Paris
  - Centre Hospitalier Universitaire Poitiers, Poitiers
  - Centre Hospitalier Quimper, Quimper
  - AUB Santé - Rennes, Rennes
  - Centre Hospitalier Universitaire Rennes, Rennes
  - Centre Hospitalier Universitaire Rouen, Rouen
  - Centre Hospitalier Saint Brieuc, Saint-Brieuc
  - Centre Hospitalier Universitaire Saint Etienne, Saint-Etienne
  - Centre Hospitalier Saint-Nazaire, Saint-Nazaire
  - Centre Hospitalier Alpes Léman, Sallanches
  - Centre Hospitalier Saint-Malo, St-Malo
  - Centre Hospitalier Universitaire Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - Clinique Saint Exupéry, Toulouse
  - CHRU Bretonneau, Tours
  - Centre Hospitalier Valenciennes, Valenciennes
  - Centre Hospitalier Bretagne Atlantique, Vannes